CLINICAL TRIAL: NCT01687582
Title: Clinical and Histopathological Effect of GLP-1 Analogs on Psoriasis in Type 2 Diabetic Patients
Brief Title: Effect of GLP-1 Analogs on Psoriasis in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-DIAB-02
Record Dates: First submitted 2012-09-11; First posted 2012-09-19 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes; Psoriasis
Keywords: type 2 diabetes; psoriasis; exenatide; liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Psoriasis | interventions — Liraglutide; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GLP-1 analog (Experimental): Liraglutide, 0.6 to 1.8 mg per day or Exenatide, 5 to 10 µg twice a day.
  Interventions: Drug: GLP-1 analog

INTERVENTIONS:
Drug: GLP-1 analog — GLP-1 analog treatment
  Other Names: Liraglutide, Victoza or Exenatide, Byetta.

SUMMARY:
The aim of the study is to evaluate after 4 to 6 months the effects of a GLP-1 analog treatment on psoriatic skin lesions in patients with type 2 diabetes.

DETAILED DESCRIPTION:
The objective of this study is to analyse short and medium-term efficacy on clinical, immunological and histopathological parameters of a GLP-1 receptor agonist on moderate to severe psoriasis plaques in a group of patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients treated with oral anti-hyperglycaemic agents and/or insulin and presenting stable psoriasis plaques for at least one year, which failed to respond to previous systemic and/or topical treatments.

Exclusion Criteria:

* Type 1 diabetes
* Secondary diabetes
* Liver, renal or pancreatic disease
* Previous treatment with GLP-1 agonist or DPP-4 inhibitors agents

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Improvement of PASI score | 4 to 6 months

SECONDARY OUTCOMES:
Evolution of BMI (body mass index) | 4 to 6 months
  number of patients with weight loss
Evolution of immunological data | 4 to 6 months
  cytokines and T cells
Evolution of histopathological data | 4 to 6 months
  thickness, dermis infiltrate in skin plaques and in control areas
Evolution of glycaemic control | 4 to 6 months
  HbA1c
Evolution of routine laboratory measures | 4 to 6 months
  number of participants with biological adverse effects (pancreatitis enzymes)
Evolution of BMI | 4 to 6 months
  weight

CONTACTS AND LOCATIONS:
Overall Officials: Martin Buysschaert, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Background] Buysschaert M, Tennstedt D, Preumont V. Improvement of psoriasis during exenatide treatment in a patient with diabetes. Diabetes Metab. 2012 Feb;38(1):86-8. doi: 10.1016/j.diabet.2011.11.004. Epub 2012 Jan 9. PMID 22227407
- [Background] Hogan AE, Tobin AM, Ahern T, Corrigan MA, Gaoatswe G, Jackson R, O'Reilly V, Lynch L, Doherty DG, Moynagh PN, Kirby B, O'Connell J, O'Shea D. Glucagon-like peptide-1 (GLP-1) and the regulation of human invariant natural killer T cells: lessons from obesity, diabetes and psoriasis. Diabetologia. 2011 Nov;54(11):2745-54. doi: 10.1007/s00125-011-2232-3. Epub 2011 Jul 9. PMID 21744074